CLINICAL TRIAL: NCT00899678
Title: A Phase 2, Open-label, Multicenter Study to Assess the Safety and Efficacy of Certolizumab Pegol in Children and Adolescents With Active Crohn's Disease (NURTURE Study)
Brief Title: The Use of Certolizumab Pegol for Treatment of Active Crohn's Disease in Children and Adolescents
Acronym: NURTURE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: higher than projected discontinuation rate during Maintenance Phase
Sponsor: UCB Celltech (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C87035; 2014-004381-24 (EudraCT Number)
Expanded Access: NCT03559660 (No longer available)
Record Dates: First submitted 2009-04-29; First posted 2009-05-12 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2015-03

CONDITIONS: Crohn's Disease
Keywords: Certolizumab Pegol; Cimzia ®; Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance High-Dose (Active Comparator): Maintenance High-Dose group: 400 mg Certolizumab Pegol for subjects ≥ 40 kg or 200 mg Certolizumab Pegol for subjects 20 to < 40 kg
  Interventions: Drug: Certolizumab Pegol
- Maintenance Low-Dose (Active Comparator): Maintenance Low-Dose group: 200 mg Certolizumab Pegol for subjects ≥ 40 kg or 100 mg Certolizumab Pegol for subjects 20 to < 40 kg
  Interventions: Drug: Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab Pegol — 400 mg administered subcutaneously at once every 4 weeks for subjects ≥ 40 kg or 200 mg for subjects 20 to < 40 kg
  *prior to this dosing regimen, subjects will undergo an induction of Certolizumab Pegol administered subcutaneously every 2 weeks (total 3 injections) at of either 400 mg for subjects ≥ 40 kg or 200 mg for subjects 20 to < 40 kg
  Other Names: Cimzia; CDP870
  Arms: Maintenance High-Dose
Drug: Certolizumab Pegol — 200 mg administered subcutaneously at once every 4 weeks for subjects ≥ 40 kg or 200 mg for subjects 20 to < 40 kg
  *prior to this dosing regimen, subjects will undergo an induction of Certolizumab Pegol administered subcutaneously every 2 weeks (total 3 injections) at of either 400 mg for subjects ≥ 40 kg or 200 mg for subjects 20 to < 40 kg
  Other Names: Cimzia; CDP870
  Arms: Maintenance Low-Dose

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, pharmacokinetics, and immunogenicity of certolizumab pegol treatment in pediatric subjects, aged 6 to 17, with moderately to severely active Crohn's disease. The target enrollment is 160 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with active Crohn's Disease (CD) confirmed 3 months prior to Screening
* Subjects with a Pediatric Crohn's Disease Activity Index (PCDAI) score of > 30 at Week 0
* Subjects between the ages of 6 and 17, inclusive, prior to baseline dosing
* Subjects must weigh > 20 kg (44 lbs)
* Subjects must have normal Electrocardiogram (ECG) or no medically relevant abnormalities as assessed by the investigator
* Subjects must meet Tuberculosis (TB) screening criteria
* Subjects taking corticosteroids, antibiotics and analgesics must have stable dosing, as defined, for one week

Exclusion Criteria:

* Subjects who score > 5 on the perirectal disease item of the PCDAI at Baseline
* Subjects who have had an active enterocutaneous fistulae within 3 months prior to Baseline
* Subjects with non-enterocutaneous fistulae, signs or symptoms of bowel obstruction or short bowel syndrome
* Subjects with a functional colostomy or ileostomy
* Subjects who have had surgical bowel resection within 6 months prior to Baseline or who may be planning any resection while enrolled in the study
* Subjects with clinical suspicion of intraabdominal abscesses
* Subjects with a positive stool result for enteric pathogens and/or parasites
* Subject has received any investigational biological therapies (within or outside a clinical trial) within 12 weeks prior to Screening or has been dosed in any clinical trial using non biological therapies within 4 weeks prior to Screening
* Subjects who have lost response to another Tumor Necrosis Factor (TNF) agent
* Subjects may not use another TNF agent within 12 weeks of Screening Visit
* Subjects with any prior exposure to natalizumab
* Subjects who have received mycophenolate or thalidomide within 4 weeks prior to Screening
* Subjects who have received cyclosporin or tacrolimus within 6 months prior to Screening
* Subjects who have received parenteral corticosteroids within 2 weeks prior to Screening
* Subjects who have received corticosteroids or corticotrophins for indications other than CD within 2 weeks of Screening
* Subject has a current or recent history (within 6 months prior to Screening) of significant and severe renal, hepatic, hematological, gastrointestinal (other than CD), endocrine, pulmonary, cardiac, neurological, or cerebral disease including blood dyscrasia (eg, pancytopenia, aplastic anemia), demyelinating disease (eg, multiple sclerosis, myelitis, optic neuritis), or ischemic heart disease
* Subjects with a current sign or symptom indicating recent or chronic infections (including herpes zoster)
* Subject has negative test for Immunoglobulin G (IgG) against Varicella zoster (chicken pox)
* Subjects who have not completed their primary vaccination series, or are planning to have a live vaccine administered during the study period or up to 3 months after last dose of study drug
* Subject has a history of TB or a positive chest x-ray suggestive of TB
* Subjects with known concurrent viral hepatitis or Acquired Immune Deficiency Syndrome (AIDS) or known Human Immunodeficiency Virus (HIV) infection
* Subjects with concurrent malignancy or history of malignancy, excluding treated squamous cell carcinoma of the skin
* Subject has concurrent bowel dysplasia or a history of bowel dysplasia in the 5 years prior to Screening
* Subjects with a history lymphoproliferative disorder including lymphoma or signs and symptoms suggestive of lymphoma at any time

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2009-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (35):
- United States (24):
  - Phoenix, Arizona
  - Los Angeles, California
  - Orange, California
  - San Francisco, California
  - Aurora, Colorado
  - Hartford, Connecticut
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Rochester, Minnesota
  - Morristown, New Jersey
  - New Hyde Park, New York
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Australia (3):
  - Randwick, New South Wales
  - Herston, Queensland
  - Parkville, Victoria
- Canada (6):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
- New Zealand (2):
  - Grafton, Auckland
  - Christchurch, Canterbury

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Participant Flow refers to the Safety Set (SS) population. The Safety Population includes all subjects enrolled who received at least 1 injection of study treatment.
Pre-assignment Details: During an Induction Period (Weeks 0 to 6), subjects were administered Certolizumab Pegol (CZP) subcutaneously every 2 weeks (Q2W). Subjects who showed a clinical response at Week 6 were randomized in a 1:1 ratio to one of 2 dose groups.
  Subjects who did not respond at Week 6 were withdrawn from the study.
Groups:
- Induction Only: Induction Only is the period between the Week 0 dose and prior to first maintenance dose (Week 8). Induction Only includes all subjects who received a dose during the Induction Period but did not receive any treatment during the Maintenance Period. During the Induction Period (Weeks 0 to 6), subjects were administered Certolizumab Pegol (CZP) subcutaneously every 2 weeks (Q2W) (for a total of 3 administrations of drug) at a dose of either:
  * 400 mg for subjects ≥ 40 kg
  * 200 mg for subjects 20 to < 40 kg
- Maintenance Low-Dose: Maintenance Low-Dose group*: 200 mg Certolizumab Pegol once every 4 weeks for subjects ≥ 40 kg or 100 mg Certolizumab Pegol once every 4 weeks for subjects 20 to < 40 kg
  *prior to this dosing regimen, subjects underwent an induction of Certolizumab Pegol administered subcutaneously every 2 weeks (total 3 injections) at of either 400 mg for subjects ≥ 40 kg or 200 mg for subjects 20 to < 40 kg
- Maintenance High-Dose: Maintenance High-Dose group*: 400 mg Certolizumab Pegol once every 4 weeks for subjects ≥ 40 kg or 200 mg Certolizumab Pegol once every 4 weeks for subjects 20 to < 40 kg
  *prior to this dosing regimen, subjects underwent an induction of Certolizumab Pegol administered subcutaneously every 2 weeks (total 3 injections) at of either 400 mg for subjects ≥ 40 kg or 200 mg for subjects 20 to < 40 kg
Period: Induction Period (Weeks 0 to 6)
Arm/Group | Induction Only | Maintenance Low-Dose | Maintenance High-Dose
Started | 27 (Induction only includes subjects that discontinued before Maintenance Period.) | 37 | 35
Completed | 2 (2 subjects completed the Induction Phase, but discontinued prior to receiving any Maintenance doses.) | 37 | 35
Not Completed | 25 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0
Not completed — Lack of Efficacy | 17 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Other reason | 1 | 0 | 0
Period: Maintenance Period (Weeks 8 to 62)
Arm/Group | Induction Only | Maintenance Low-Dose | Maintenance High-Dose
Started | 0 (Induction only includes subjects that discontinued before Maintenance Period.) | 37 | 35
Completed | 0 | 12 | 7
Not Completed | 0 | 25 | 28
Not completed — Adverse Event | 0 | 10 | 5
Not completed — Lack of Efficacy | 0 | 11 | 18
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Other reason | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Baseline characteristics refer to the Safety Set (SS) population. The Safety Population includes all subjects enrolled who received at least 1 injection of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction Only | Maintenance Low-Dose | Maintenance High-Dose | Total
Number analyzed (Participants) | 27 | 37 | 35 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (2.67) | 13.2 (2.41) | 13.4 (2.46) | 13.4 (2.48)
Age, Customized [Number; unit: participants]
  6-11 years | 6 | 9 | 8 | 23
  12-17 years | 21 | 28 | 27 | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 21 | 41
  Male | 17 | 27 | 14 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian / Alaskan Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Black | 3 | 3 | 8 | 14
  Native Hawaiian or other Pacific islander | 0 | 0 | 0 | 0
  White | 22 | 32 | 27 | 81
  Other / Mixed | 1 | 2 | 0 | 3
Weight [Mean (Standard Deviation); unit: kilogram] | 46.50 (12.565) | 45.67 (14.638) | 50.35 (18.569) | 47.55 (15.642)
Height [Mean (Standard Deviation); unit: centimeter] | 157.46 (13.841) | 155.32 (13.589) | 157.22 (13.320) | 156.57 (13.460)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter] | 18.39 (2.504) | 18.51 (3.531) | 19.79 (4.897) | 18.93 (3.869)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meter] | 1.42 (0.250) | 1.39 (0.272) | 1.47 (0.319) | 1.43 (0.283)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects in Clinical Remission at Week 62
Description: Clinical remission is defined as a Pediatric Crohn's Disease Activity Index (PCDAI) score ≤ 10.
  The Pediatric Crohn's Disease Activity Index (PCDAI) consists of 4 domains (laboratory, height/weight, examination, and history) with several assessments that are converted into a PCDAI score which can range from 0 to 100 points, with a higher score indicating more severe disease activity.
Time Frame: Week 62
Population: Full Analysis Set (FAS) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Low-Dose | Maintenance High-Dose
Number analyzed (Participants) | 37 | 35
percentage of participants | 24.3 [10.5 to 38.1] | 17.1 [4.7 to 29.6]

2. Secondary Outcome: Absolute Pediatric Crohn's Disease Activity Index (PCDAI) Scores at Week 62
Description: The Pediatric Crohn's Disease Activity Index (PCDAI) consists of 4 domains (laboratory, height/weight, examination, and history) with several assessments that are converted into a PCDAI score which can range from 0 to 100 points, with a higher score indicating more severe disease activity.
Time Frame: Week 62
Population: Full Analysis Set (FAS) population. At the start of the Maintenance Period, the FAS had 37 subjects in the Low-Dose group and 35 subjects in the High-Dose group. However, at Week 62, there were only 11 subjects in the Low-Dose group and 7 subjects in the High-Dose group with valid Pediatric Crohn's Disease Activity Index (PCDAI) scores.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Maintenance Low-Dose | Maintenance High-Dose
Number analyzed (Participants) | 11 | 7
Score on a scale | 8.18 (6.900) | 7.14 (7.830)

3. Secondary Outcome: Change in Pediatric Crohn's Disease Activity Index (PCDAI) Scores From Week 0 to the End of the Study (Week 62)
Description: The Pediatric Crohn's Disease Activity Index (PCDAI) consists of 4 domains (laboratory, height/weight, examination, and history) with several assessments that are converted into a PCDAI score which can range from 0 to 100 points, with a higher score indicating more severe disease activity.
  A negative value in change from Baseline indicates an improvement from Baseline to Week 62.
Time Frame: From Week 0 to Week 62
Population: Full Analysis Set (FAS) population. At the start of the Maintenance Period, the FAS had 37 subjects in the Low-Dose group and 35 subjects in the High- Dose group. However, at Week 62, there were only 11 subjects in the Low-Dose group and 7 subjects in the High-Dose group with valid Pediatric Crohn's Disease Activity Index (PCDAI) scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Low-Dose | Maintenance High-Dose
Number analyzed (Participants) | 11 | 7
units on a scale | -29.77 (8.097) | -27.14 (5.669)

4. Secondary Outcome: Percentage of Subjects Achieving Clinical Response From Week 0 to the End of the Study (Week 62)
Description: Clinical response is defined as a decrease from Week 0 in Pediatric Crohn's Disease Activity Index (PCDAI) score of ≥ 15 points and a total PCDAI score ≤ 30 points.
  The Pediatric Crohn's Disease Activity Index (PCDAI) consists of 4 domains (laboratory, height/weight, examination, and history) with several assessments that are converted into a PCDAI score which can range from 0 to 100 points, with a higher score indicating more severe disease activity.
Time Frame: From Week 0 to Week 62
Population: Full Analysis Set (FAS) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Low-Dose | Maintenance High-Dose
Number analyzed (Participants) | 37 | 35
percentage of participants | 29.7 [15.0 to 44.5] | 20.0 [6.7 to 33.3]

5. Secondary Outcome: C-Reactive Protein (CRP) Levels at Week 62
Description: The C-Reactive Protein (CRP) is a considered marker of inflammation in subjects with Crohn's Disease (CD)
Time Frame: Week 62
Population: Full Analysis Set (FAS) population. At the start of the Maintenance Period, the FAS had 37 subjects in the Low-Dose group and 35 subjects in the High- Dose group. However, at Week 62, there were only 11 subjects in the Low-Dose group and 7 subjects in the High-Dose group with valid C-Reactive Protein (CRP) levels.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Maintenance Low-Dose | Maintenance High-Dose
Number analyzed (Participants) | 11 | 7
mg/L | 7.2 [2.5 to 20.7] | 5.8 [2.1 to 15.7]

6. Secondary Outcome: Change in C-Reactive Protein (CRP) Levels From Week 0 to the End of the Study (Week 62)
Description: The C-Reactive Protein (CRP) is a considered marker of inflammation in subjects with Crohn's Disease (CD).
  Changes from Baseline in CRP levels are expressed as a ratio with the value measured at Baseline as the denominator.
Time Frame: From Week 0 to Week 62
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Maintenance Low-Dose | Maintenance High-Dose
Number analyzed (Participants) | 11 | 7
ratio | 0.49 [0.17 to 1.41] | 1.84 [0.27 to 12.71]

7. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) at Week 62
Description: The Erythrocyte Sedimentation Rate (ESR) is a considered biomarker of inflammation in subjects with Crohn's Disease (CD).
Time Frame: Week 62
Population: Full Analysis Set (FAS) population. At the start of the Maintenance Period, the FAS had 37 subjects in the Low-Dose group and 35 subjects in the High- Dose group. However, at Week 62, there were only 12 subjects in the Low-Dose group and 7 subjects in the High-Dose group with a valid Erythrocyte Sedimentation Rate (ESR).
Measure: Geometric Mean (95% Confidence Interval); unit: mm/h
Arm/Group | Maintenance Low-Dose | Maintenance High-Dose
Number analyzed (Participants) | 12 | 7
mm/h | 20.9 [11.8 to 37.2] | 25.2 [12.3 to 51.7]

8. Secondary Outcome: Change in Erythrocyte Sedimentation Rate (ESR) From Week 0 to the End of the Study (Week 62)
Description: The Erythrocyte Sedimentation Rate (ESR) is a considered biomarker of inflammation in subjects with Crohn's Disease (CD).
  Changes from Baseline in CRP levels are expressed as a ratio with the value measured at baseline as the denominator.
Time Frame: From Week 0 to Week 62
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Maintenance Low-Dose | Maintenance High-Dose
Number analyzed (Participants) | 12 | 7
ratio | 0.57 [0.31 to 1.04] | 1.08 [0.39 to 3.02]

9. Secondary Outcome: Change in Growth Scores (Tanner Stage [Assessing Puberty]) From Week 0 to the End of the Study (Week 62)
Description: The Tanner stage is an assessment of developmental stage on external genitalia and pubic hair (boys), and on breast and pubic hair (girls). Values range from 1 to 5 where a higher number indicates more development.
Time Frame: From Week 0 to Week 62
Population: Full Analysis Analysis (FAS) population. At the start of the Maintenance Period, the FAS had 37 subjects in the Low-Dose group and 35 subjects in the High- Dose group. However, at Week 62, there were only 10 subjects in the Low-Dose group and 7 subjects in the High-Dose group with valid Growth scores.
Measure: Number; unit: participants
Arm/Group | Maintenance Low-Dose | Maintenance High-Dose
Number analyzed (Participants) | 10 | 7
participants
  Increase from Stage I to Stage II | 2 | 0
  Increase from Stage I to Stage III | 1 | 1
  Increase from Stage II to Stage III | 0 | 1
  Increase from Stage III to Stage IV | 2 | 0
  Increase from Stage IV to Stage V | 0 | 1
  Decrease from Stage IV to Stage III | 1 | 1
  Subjects remained in Stage I | 0 | 1
  Subjects remained in Stage III | 0 | 2
  Subjects remained in Stage IV | 1 | 0
  Subjects remained in Stage V | 3 | 0

10. Secondary Outcome: Percentage of Subjects Who Initiated Steroid Tapering
Description: Subjects receiving corticosteroids at Screening may start a defined tapering schedule between Weeks 2 and 8. Corticosteroid tapering must start at the latest by Week 8. Corticosteroid doses are tapered at different rates depending on the subject's dose.
Time Frame: From Week 2 up to Week 8
Population: Full Analysis Set (FAS) population. There were only 21 subjects in the Low-Dose group and 20 subjects in the High-Dose group who took steroids during the Maintenance Period.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Maintenance Low-Dose | Maintenance High-Dose
Number analyzed (Participants) | 21 | 20
percentage of subjects | 71.4 [52.1 to 90.8] | 65.0 [44.1 to 85.9]

11. Secondary Outcome: Percentage of Subjects in Corticosteroid-free Remission at the End of the Study
Description: Corticosteroid use at end of study is defined as 84 days past the last dose of study medication. Remission is assessed at the last visit where Pediatric Crohn's Disease Activity index (PCDAI) data is available.
Time Frame: Last/Withdrawal Visit (up to Week 62)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | Maintenance Low-Dose | Maintenance High-Dose
Number analyzed (Participants) | 21 | 20
percentage of paticipants | 23.8 [5.6 to 42.0] | 15.0 [0.0 to 30.6]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over 68 weeks (from Week -6 to Week 62).
Description: Adverse Events (AEs) refer to the Safety Set (SS) population. All subjects in the Safety Population (n=99) participated in the Induction Period. There were 27 subjects who did not continue into the Maintenance Period.
Groups:
- Induction Period: Induction Only is the period between the Week 0 dose and prior to first maintenance dose (Week 8). Induction Only includes all subjects who received a dose during the Induction Period but did not receive any treatment during the Maintenance Period. During the Induction Period (Weeks 0 to 6), subjects were administered Certolizumab Pegol (CZP) subcutaneously every 2 weeks (Q2W) (for a total of 3 administrations of drug) at a dose of either:
  * 400 mg for subjects ≥ 40 kg
  * 200 mg for subjects 20 to < 40 kg
- Overall Study: Overall Study comprises Induction Period and Maintenance Period (Week -6 to Week 62).
Arm/Group | Induction Period | Maintenance Low-Dose | Maintenance High-Dose | Overall Study
Serious Adverse Events (participants affected / at risk) | 6/99 | 4/37 | 4/35 | 14/99
Other Adverse Events (participants affected / at risk) | 59/99 | 28/37 | 27/35 | 78/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period (N=99) | Maintenance Low-Dose (N=37) | Maintenance High-Dose (N=35) | Overall Study (N=99)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period (N=99) | Maintenance Low-Dose (N=37) | Maintenance High-Dose (N=35) | Overall Study (N=99)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (4) | 4 (4) | 10 (12)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 5 (5) | 2 (3) | 9 (12)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 7 (7)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 5 (7) | 7 (8) | 12 (15)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 3 (5) | 3 (7) | 12 (19)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 5 (6)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 8 (8)
Nausea (Gastrointestinal disorders) | 6 (8) | 3 (3) | 2 (2) | 10 (13)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2) | 5 (6)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (4)
Vomiting (Gastrointestinal disorders) | 6 (7) | 3 (3) | 6 (10) | 13 (20)
Fatigue (General disorders) | 3 (3) | 3 (4) | 0 (0) | 6 (7)
Injection site pain (General disorders) | 22 (55) | 4 (17) | 6 (36) | 22 (108)
Pyrexia (General disorders) | 9 (15) | 6 (7) | 9 (9) | 20 (31)
Ear infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 2 (3) | 6 (7)
Nasopharyngitis (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 8 (8)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 8 (9) | 2 (2) | 10 (11)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Viral infection (Infections and infestations) | 2 (3) | 4 (4) | 3 (5) | 9 (12)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Weight decreased (Investigations) | 2 (2) | 2 (2) | 1 (3) | 4 (7)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 1 (1) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (4) | 2 (2) | 12 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 9 (12) | 4 (10) | 3 (4) | 12 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 2 (5) | 8 (13)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 2 (2) | 8 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (6) | 0 (0) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days